CLINICAL TRIAL: NCT05339308
Title: Effects of Magnesium Oil Application on the Muscle Contractile Properties
Acronym: MG-MCP2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Armin Paravlic, Principal Investigator, University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MG-MCP2022
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Magnesium; Skeletal Muscle Contraction Properties
Keywords: Tensiomyography; Skeletal Muscle; Contractile Properties
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will not be informed about the actual study purpose, while the main investigator will be blinded to the EXP or CON oil administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Magnesium oil application
  Interventions: Other: Magnesium oil (BetterYou) dermal application
- Control (Placebo Comparator): Natural mineral-free oil application
  Interventions: Other: Placebo Control

INTERVENTIONS:
Other: Magnesium oil (BetterYou) dermal application — 10 sprays (200 mg) of magnesium oil (BetterYou) will be applied to skin covering knee extensor muscles. The magnesium oil will be applied only once
  Arms: Experimental
Other: Placebo Control — Natural mineral-free oil (10 sprays) will be applied as the control condition. This will be done only once
  Other Names: CONTROL
  Arms: Control

SUMMARY:
This study will aim to investigate the effects of magnesium oil administration on skeletal muscle contractile properties.

DETAILED DESCRIPTION:
Aim: This study will aim to investigate the effects of magnesium oil administration on skeletal muscle contractile properties (SMcp).

Design: Randomized controlled study

Participants: For this purpose, investigators will recruit 40 recreationally active and healthy adults of both sexes (18-35 years of age).

Methods: The experimental leg (EXP) will receive the 10 sprays of magnesium oil (20 mg per spray) that will be topically applied to the skin covering the knee extensor muscles, whereas the control leg (CON) will receive 10 sprays of natural mineral-free oil. The vastus lateralis SMcp will be measured by using a tensiomyography (TMG) device before application (PRE) and after 10 (POST10), 20 (POST20), 30 (POST30), 40 (POST40), and 50 (POST50) minutes of application onset, respectively.

ELIGIBILITY:
Inclusion Criteria:

* healthy, recreationally active adults, no history of neuromuscular and musculoskeletal diseases

Exclusion Criteria:

* if some of the criteria are not met

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Contractile Properties | 75 minutes
  Skeletal muscle contractile properties will be measured by using tensiomyography device

CONTACTS AND LOCATIONS:
Overall Officials: Armin Paravlic, PhD, Principal Investigator — Faculty of Sport
Locations (2):
- Masaryk University, Brno, Czechia
- Faculty of Sport, Ljubljana, Slovenia, Slovenia

IPD SHARING:
Plan to Share IPD: No